CLINICAL TRIAL: NCT03554161
Title: Efficacy and Safety of Tocilizumab in the Treatment of Refractory Uveitis in Patients With Behcet's Disease
Brief Title: Tocilizumab for the Treatment of Refractory Behcet's Uveitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on its primary and secondary outcome measures in three consecutive patients.
Sponsor: Wenjie Zheng (Other)
Responsible Party: Sponsor-Investigator, Wenjie Zheng, Professor， Department of Rheumatology, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCZ-BDU-PUMCH
Record Dates: First submitted 2018-04-21; First posted 2018-06-13 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Behcet Syndrome; Uveitis
Keywords: Tocilizumab; Refractory uveitis
MeSH Terms: conditions — Behcet Syndrome; Uveitis | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Tocilizumab is approved for the treatment of several inflammatory disease, this study tends to evaluate the response to TCZ in refractory BDU, thus it is a self-control study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tocilizumab for refractory BDU (Experimental): This study is a self-control study and all the participants will be enrolled in the interventional arm.
  Interventions: Biological: Tocilizumab (TCZ)

INTERVENTIONS:
Biological: Tocilizumab (TCZ) — Patients with refractory BD associated uveitis will receive Tocilizumab therapy, the efficacy and corticosteroids-tapering effects will be evaluated.

SUMMARY:
The aim of this single-center prospective study is to evaluate the efficacy and safety of Tocilizumab (TCZ), humanized monoclonal antibody against IL-6receptor, in the treatment of refractory Uveitis of Behçet's disease (BDU), to verify its effects on decreasing the dose of cortical steroids, and to determine whether it can reduce BDU recurrence.

DETAILED DESCRIPTION:
Uveitis of Behçet's disease (BDU) is the most common form of ocular manifestations, which is also the leading cause of irreversible visual impairment. The aim of the study is to Improve treatment strategy of the disease as well as to reduce blindness.

Tocilizumab (TCZ) is a humanized antibody against IL-6 receptor, clinical trials on non-infectious uveitis and retrospective study on BDU has obtained expected results.

This single-center prospective study is to evaluate the efficacy and safety of TCZ in the treatment of refractory BDU, to verify its effects on decreasing the dose of corticosteroids, and to determine whether it can reduce BDU recurrence.The investigators aim to enroll nine refractory BDU patients with acute onset uveitis, with difficulty tapering corticosteroids while being treated with at least one of the commonly used immunosuppressants. All participants will receive TCZ , oral corticosteroids and immunosuppressants will remain unchanged, intraocular injection will be avoided. During monthly follow-up, the investigators will measure and record intraocular inflammation status，as well as extraocular manifestations and the acute-phase reactants. The participants will continue to receive TCZ for six months, the primary end point is the efficacy four weeks after first dose of TCZ, secondary end points other than intraocular inflammation will be achieved on each follow-up visit, as quality of life improvements, side effects, recurrence of uveitis, and corticosteroids-tapering effects.

On statistical analysis, the self-control treatment efficiency and recurrence rate difference will be determined using T-test of paired samples at a significance level of 0.05(2-sided).

To ensure the interest of the participants, the study has been reviewed by the PUMCH ethics committee, and drug clinical research liability insurance was prepared.

ELIGIBILITY:
Inclusion Criteria:

* All participants fulfill the the proposed International Criteria for BD, either ISG criteria(1990) or ICBD criteria(2013).
* All participants present with refractory BDU , acute onset uveitis, either posterior segment involvement or panuveitis, with difficulty tapering corticosteroids while being treated with at least one of the commonly used immunosuppressants, without severe extraocular manifestations.

Exclusion Criteria:

* Patients with impaired hepatic and renal function, other severe ocular diseases, active tuberculosis, viral hepatitis, malignancy, pregnancy will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Tocilizumab on BD Uveitis | four weeks
  Remission or deterioration of uveitis，based on intraocular inflammation evaluation

SECONDARY OUTCOMES:
Intraocular inflammation evaluation BOS24 index | each follow-up visit / every four weeks, up to six months
  Visual acuity, anterior chamber cells, vitreous opacities, retinal inflammation, macular thickness, etc.
Corticosteroid-tapering effects | six months
  Whether corticosteroid dosage could be tapered to minimum dose.
Reduction of uveitis recurrence | each follow-up visit / every four weeks, up to six months
  Differences of recurrence between before and after treatment
Severity of uveitis on recurrence | each follow-up visit / every four weeks, up to six months
  Differences of severity of recurrence between before and after treatment
Improvement of quality of life | each follow-up visit / every four weeks, up to six months
  Record quality of life on questionnaire: BDCAF
Improvement of quality of life | each follow-up visit / every four weeks, up to six months
  Record quality of life on questionnaire: SF-36
Side effects of treatment | each follow-up visit / every four weeks, up to six months
  Record any side effects during intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Zheng, M.D., Principal Investigator — Department of Rheumatology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Atienza-Mateo B, Calvo-Rio V, Beltran E, Martinez-Costa L, Valls-Pascual E, Hernandez-Garfella M, Atanes A, Cordero-Coma M, Miquel Nolla J, Carrasco-Cubero C, Loricera J, Gonzalez-Vela MC, Vegas-Revenga N, Fernandez-Diaz C, Demetrio-Pablo R, Dominguez-Casas LC, Luis Martin-Varillas J, Palmou-Fontana N, Hernandez JL, Gonzalez-Gay MA, Blanco R. Anti-interleukin 6 receptor tocilizumab in refractory uveitis associated with Behcet's disease: multicentre retrospective study. Rheumatology (Oxford). 2018 May 1;57(5):856-864. doi: 10.1093/rheumatology/kex480. PMID 29471416
- [Result] Lopalco G, Fabiani C, Sota J, Lucherini OM, Tosi GM, Frediani B, Iannone F, Galeazzi M, Franceschini R, Rigante D, Cantarini L. IL-6 blockade in the management of non-infectious uveitis. Clin Rheumatol. 2017 Jul;36(7):1459-1469. doi: 10.1007/s10067-017-3672-z. Epub 2017 May 20. PMID 28528519
- See also: Springerlink — http://link.springer.com/article/10.1007%2Fs10067-017-3672-z